CLINICAL TRIAL: NCT05991505
Title: Effect of Distance Physical Exercise on Mobility and Sleep Quality of Hypertensive Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nereida Kilza da Costa Lima, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5174
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Aging Well; Training Group, Sensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Control (No Intervention): Volunteers with no physical activity during 10 weeks
- 2 - Training (Active Comparator): Volunteers with supervised home physical activity, twice a week, during 10 weeks
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Multimodal exercises twice a week
  Arms: 2 - Training

SUMMARY:
The objective of the present study was to verify the impact of physical exercise at a distance (EFAD) on the level of mobility and quality of sleep of hypertensive elderly women. To this end, hypertensive elderly women under drug treatment aged between 60 and 79 years old age, without orthopedic limitations and/or cardiovascular complaints were assessed using questionnaires, functional tests, sleep scale classification and use of actigraphy for 7 days. Afterwards, they were randomized into 2 groups, control and EFAD, with synchronous training online 2x/week and by recorded class 1x/week. Reassessments were made after 10 weeks.

DETAILED DESCRIPTION:
Weight was checked using an OMRON model HBF-214 scale and height was checked using a 2-meter Slim Fit compact stadiometer, after which the body mass index (BMI) was calculated. All procedures took approximately 35 minutes, supervised by the researcher in charge. The researcher used personal protective equipment, such as an N95 mask and frequent use of alcohol gel on hands and surfaces. All participants and researchers involved in the study were vaccinated against SARS COV-2 according to the health status of the study period.

Physical tests were performed after measuring blood pressure (BP) with values equal to or less than 160x100 mmHg. The Timed Up and Go (TUG) test was performed to assess the participants' mobility and risk of falling. Studies show a greater risk of falling with times above 20 seconds. After the TUG, the gait speed test was performed, as it is an important predictor of cardiovascular health. In this test, a speed equal to or greater than 0.89 meters per second is expected in elderly people with preserved capacity.

Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire . There are 19 questions grouped into seven categories: subjective sleep quality; sleep latency; nocturnal sleep duration; sleep effectiveness; sleep disorders; sleeping pills; daytime sleepiness. Each category is scored from 0 to 3, allowing a total sum of 0 to 21. Values above 9 in the total sum indicate poor sleep quality. This questionnaire is validated and widely used. In addition to this questionnaire, the Epworth sleepiness scale was used, containing 8 questions with scores from 0 to 3 points in each situation, with abnormal sleepiness classification above 9 points.

Subjects were also assessed for sleep quality with actigraphy. The ActTrust device, Condor Instruments - Brazil was used. The device was placed on the participant's non-dominant wrist. Participants' activities were monitored for a period of 7 days (24 hours), allowing for an objective analysis of sleep quality. At the end of this period, a new home visit was carried out to remove the actigraph and the information was transferred through a USB interface and specific software that performed the data analysis.

ELIGIBILITY:
Inclusion Criteria: hypertensive women in regular use of medication prescribed for high blood pressure, physically active, and with basic knowledge to use smartphones, tablets, with internet access and able to understand and answer the survey questionnaires.

-

Exclusion Criteria:orthopedic limitations, cardiovascular complaints or limitation for performing basic movements

-

Ages: 60 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of sleep | 1
  Quality of sleep evaluated by actigraphy and Pittsburgh Sleep Quality Index

SECONDARY OUTCOMES:
Mobility | 2
  Mobility evaluated by Timed up and Go Test and walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Moriguti, MD, PhD, Study Chair — Ribeirão Preto Medical School - USP
Locations (1):
- Clinics Hospital, Ribeirão Preto Medical School, University of São Paulo, Ribeirão Preto, São Paulo, Brazil